CLINICAL TRIAL: NCT02768246
Title: Comparison of the Efficacy of a Bag-Valve-Guedel Adaptor to the Commonly Used Face Mask in Healthy Bearded Volunteers
Brief Title: Comparison of Bag-Valve-Guedel Adaptor to Common Face Mask for the Ventilation of Bearded Men
Acronym: BVGA01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Lilach Gavish, Study Director, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0051-16-HMO
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Pre-hospital Ventilation
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Begin with BVGA (Active Comparator): The volunteers will be asked to breathe 5 minutes of room air through the BVGA, followed by, 5 minutes 100% oxygen, and 5 minutes room air again. This will be followed by 5 minutes room air breathing without the BVGA. Then the same volunteers will be asked to repeat the protocol with the face mask.
  Interventions: Device: BVGA; Device: Face Mask
- Begin with Face-mask (Active Comparator): The volunteers will be asked to breathe 5 minutes of room air through the face mask, followed by, 5 minutes 100% oxygen, and 5 minutes room air again. This will be followed by 5 minutes room air breathing without the face mask. Then the same volunteers will be asked to repeat the protocol with the BVGA.
  Interventions: Device: BVGA; Device: Face Mask

INTERVENTIONS:
Device: BVGA — The BVGA enables the direct connection of a bag valve device to a guedel, eliminating the need for a face mask during ventilation
  Other Names: Bag Valve Guedel Adaptor
Device: Face Mask — Classic face mask

SUMMARY:
Ventilation of a bearded patient with the commonly used face mask has low efficiency because of difficulties to achieve a tight seal around the mouth and nose.

The purpose of this study is to evaluate the efficacy of a novel bag valve guedel adaptor (BVGA) that enables the direct connection of a bag valve device to a guedel - eliminating the need for a face mask.

DETAILED DESCRIPTION:
Ventilating a patient using a bag valve and a face mask is not easy to perform, especially for a long period of time, and mandates experience and strength by the care giver. The need for a tight seal around the mouth and nose is a major challenge especially if the patient has a beard. Nevertheless, the face mask is the only approved respiratory support that medics and other basic care givers are allowed to use in the out-of-the-hospital setting, and only physicians and paramedics are allowed to use more advanced techniques, providing a definite airways. Thus, despite its lower effectiveness, the bag valve mask technique is the most commonly used in the field

The purpose of this study is to evaluate the efficacy of a novel bag valve guedel adaptor (BVGA) that enables the direct connection of a bag valve device to a guedel - eliminating the need for a face mask.

Study Design: Prospective, randomized, controlled. The volunteers will be asked randomly assigned to breathe through the BVGA/Face mask followed by the same protocol with the Face-mask/BVGA: 5 minutes room air, 5 minutes 100% oxygen, and 5 minutes room air again. The BVGAs/face masks well be connected to a standard operating room ventilation machines, and cardiopulmonary parameters will be monitored and documented.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males more than 18 years of age.
2. 22 with beards, 3 without beards.

Exclusion Criteria:

1. Presence of facial fractures or injuries.
2. Claustrophobia.
3. Respiratory diseases.
4. Severe illness such as cardiac or neurological diseases.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
End tidal CO2 levels (EtCO2) | 30 minutes
  EtCO2 will be monitored while the volunteer breathes through the BVGA or the face mask.

SECONDARY OUTCOMES:
End tidal O2 (EtO2) | 30 minutes
  EtO2 will be monitored while the volunteer breathes through the BVGA or the face mask.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Shaylor, MD, Principal Investigator — Hadassah Medical Organization; Lilach Gavish, PhD, Study Director — Hebrew University of Jerusalem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavish L, Rittblat M, Gertz SD, Shaylor R, Weissman C, Eisenkraft A. Ventilating the Bearded: A Randomized Crossover Trial Comparing a Novel Bag-Valve-Guedel Adaptor to a Standard Mask. Mil Med. 2020 Aug 14;185(7-8):e1300-e1308. doi: 10.1093/milmed/usz378. PMID 33444455